CLINICAL TRIAL: NCT03216655
Title: Comparison of Individual and Cohort Long Distance Advising for Mental Care for Congenital Cataract Guardians
Brief Title: Individual vs Cohort Long Distance Advising for Mental Care for Congenital Cataract Guardians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CCPMOH2017-China-1
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Cataract
Keywords: congenital cataract; anxiety; guardian
MeSH Terms: conditions — Cataract; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional group (Experimental): phone call
  Interventions: Other: phone call
- new device group (Experimental): wechat group
  Interventions: Other: wechat group

INTERVENTIONS:
Other: phone call — Investigators give a regular follow-up to participants: phone call monthly
  Arms: traditional group
Other: wechat group — Investigators give a regular follow-up to participants: wechat follow up. Investigators send useful information and answer their questions monthly.
  Arms: new device group

SUMMARY:
Nowadays, doctors put mental health at a prior place and pay more attention to the psychological problems of ill kids' parents. In our research, we try to find a new modern and efficient psychological counseling mode to improve the mentality of parents and relieve their anxiety and depression. We divide guardians of parents into two groups .One group is given the traditional follow-up by regular phone call every month. The other is in a wechat group. A doctor send the useful information about kids care and answer questions of parents at regular time every month. The self-rating anxiety scale (SAS) and self-rating depression scale (SDS) scores of parents are marked before and after the long follow up.

DETAILED DESCRIPTION:
Congenital cataract (CC) is the leading cause of reversible blindness during childhood, which appears at birth or during the first decade of life. Nowadays, doctors put mental health at a prior place and pay more attention to the psychological problems of ill kids' parents. In our research, we try to find a new modern and efficient psychological counseling mode to improve the mentality of parents and relieve their anxiety and depression. We divide guardians of parents into two groups .One group is given the traditional follow-up by regular phone call every month. The other is in a wechat group. A doctor send the useful information about kids care and answer questions of parents at regular time every month. The self-rating anxiety scale (SAS) and self-rating depression scale (SDS) scores of parents are marked before and after the long follow up.

ELIGIBILITY:
Inclusion Criteria: the guardians of kids who had a surgery for congenital cataract recently

Exclusion Criteria:

have other major life hit was diagnosed of anxiety and depression before

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
similar effect | baseline
  the SAS and SDS level are same in two groups
efficient effect | baseline
  the SAS and SDS level are higher in traditional group
invalid effect | baseline
  the SAS and SDS level are lower in traditional group

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D,Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China